CLINICAL TRIAL: NCT05735093
Title: The Effect of Dcr3 Levels in Blood and Urine on Renal and Patient Prognosis in Patients With Acute Kidney Injury
Brief Title: Dcr3 Levels in Blood and Urine on Renal and Patient Prognosis in Patients With Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Betul Deniz Gozmen, Dr Betul Deniz Gozmen, Kırıkkale University
Other Study IDs: 2022/009
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury
Keywords: DcR levels, renal prognosis, patient survival, acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney diseases represent a global public health problem due to the aging of the population, the increasing prevalence of diabetes, hypertension, obesity and immune disorders. TNF-superfamily ligands are heterotrimeric transmembrane proteins with a molecular structure characterized by the presence of a TNF homology domain that binds to cysteine-rich regions of specific TNF-superfamily receptors. The tumor necrosis factor (TNF) superfamily consists of ligands and receptors that modulate adaptive immunity regulation, hematopoiesis, morphogenesis, as well as different disease states, including cancer and diabetes. DcR3 is found increased in a variety of cancer cells and various inflammatory tissues and is considered a potential biomarker to predict inflammatory disease progression and cancer metastasis. While increasing DcR3 expression may be possible to treat inflammatory diseases and enhance tissue repair, decreasing DcR3 expression may increase tumor apoptosis and suppress tumor growth in vivo. The study will be carried out with the prospective examination of patients without anuria and who developed Acute Kidney Injury or on the basis of Acute Kidney Disease on Chronic Kidney Disease. Sixty patients and 30 age- and gender matched control healthy individuals that accept enrollment in the study will be followed up by the Nephrology Department in Kırıkkale University Faculty of Medicine for 2 years. The aim of this study was to investigate the relationship between blood and urine DcR 3 levels on the effects of renal and patient prognosis in patients with Acute Kidney Injury as a predictor or an auxiliary test in prediction.

DETAILED DESCRIPTION:
Kidney diseases represent a global public health problem due to the aging of the population, the increasing prevalence of diabetes, hypertension, obesity and immune disorders. TNF-superfamily ligands are heterotrimeric transmembrane proteins with a molecular structure characterized by the presence of a TNF homology domain that binds to cysteine-rich regions of specific TNF-superfamily receptors. The tumor necrosis factor (TNF) superfamily consists of ligands and receptors that modulate adaptive immunity regulation, hematopoiesis, morphogenesis, as well as different disease states, including cancer and diabetes. DcR3 is found increased in a variety of cancer cells and various inflammatory tissues and is considered a potential biomarker to predict inflammatory disease progression and cancer metastasis. While increasing DcR3 expression may be possible to treat inflammatory diseases and enhance tissue repair, decreasing DcR3 expression may increase tumor apoptosis and suppress tumor growth in vivo. The study will be carried out with the prospective examination of patients without anuria and who developed Acute Kidney Injury or on the basis of Acute Kidney Disease on Chronic Kidney Disease. Sixty patients and 30 age- and gender matched control healthy individuals that accept enrollment in the study will be followed up by the Nephrology Department in Kırıkkale University Faculty of Medicine for 2 years. The aim of this study was to investigate the relationship between blood and urine DcR 3 levels on the effects of renal and patient prognosis in patients with Acute Kidney Injury as a predictor or an auxiliary test in prediction.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Agree to participate in the study
* Patients with previously normal kidney function and Chronic Kidney Disease patients not receiving replacement therapy
* The patient is not anuric
* Malignant and inflammatory, autoimmune disease not having a history.

Exclusion Criteria:

* Non-Acute kidney injury dialysis procedures (Intox etc.)
* Chronic kidney disease patients receiving dialysis treatment
* Renal replacement therapy was started due to acute kidney injury in an external center, patients referred to our center
* Pediatric age patients
* Malignancy
* Chronic inflammatory and autoimmune disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-90 years old Male and female Patients with acute kidney injury
Sampling Method: Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Renal Survival | 12 months
  Dobling of serum creatinine and kidney replacement therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: UCLER KISA, Prof, Study Chair — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Yahsihan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No